CLINICAL TRIAL: NCT03140514
Title: Urine CXCL10 Chemokine Monitoring Post-renal Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Urine chemokine monitoring
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Renal Transplant Rejection
Keywords: Urine chemokine monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Urine CXCL10-chemokine levels will be monitored at specific time points post-transplant. Sustained elevated levels will trigger performance of a renal allograft biopsy. Any rejection will be treated. Rejection treatment according to clinical standard-of-care
  Interventions: Drug: Rejection treatment according to clinical standard-of-care
- Control (No Intervention): Urine CXCL10-chemokine levels will be monitored at specific time points post-transplant, but the values are concealed.

INTERVENTIONS:
Drug: Rejection treatment according to clinical standard-of-care — Standard-of-care treatment is based on the severity and phenotype of biopsy-proven rejection
  Arms: Intervention

SUMMARY:
In this study investigators will investigate whether early treatment of allograft rejection, as detected by urine CXCL10-monitoring, improves outcomes in renal allograft recipients.

ELIGIBILITY:
Inclusion Criteria:

* All consenting adult (age>=18) renal allograft recipients

Exclusion Criteria:

* Human Leucocyte Antigen (HLA) -identical living donor transplantation
* Primary non-function
* Participation in immunosuppression interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Graft loss not due to death of the patient | First year post-transplant
  1-year composite outcome consisting of at least one of the primary outcomes 1 to 4
Biopsy-proven clinical acute rejection | 4-weeks up to 1-year post-transplant
  1-year composite outcome consisting of at least one of the primary outcomes 1 to 4
Subclinical T-cell mediated rejection in 1-year surveillance biopsy defined by t>0 and/or v>0 | First year post-transplant
  1-year composite outcome consisting of at least one of the primary outcomes 1 to 4
Interstitial fibrosis / tubular atrophy with inflammation (IFTA+i defined by the Mayo Clinic criteria) in 1-year surveillance biopsy | First year post-transplant
  1-year composite outcome consisting of at least one of the primary outcomes 1 to 4

SECONDARY OUTCOMES:
Efficacy assessed by microvascular inflammation at 1-year (ptc, g, c4d, cg) | First year post-transplant
  Microvascular inflammation at 1-year (ptc, g, c4d, cg)
Efficacy assessed by development of IFTA from implantation to 1-year (∆ ci, ct, cv) | First year post-transplant
  Development of IFTA from implantation to 1-year (∆ ci, ct, cv)
Efficacy assessed by number of days from transplantation to biopsy-proven clinical acute rejection | First year post-transplant
  number of days from transplantation to biopsy-proven clinical acute rejection
Efficacy assessed by Proteinuria >500mg/day at 6- and 12-months post-transplant | First year post-transplant
  Proteinuria >500mg/day at 6- and 12-months post-transplant
Safety assessed by total number of biopsies, indication for biopsy and CXCL10-triggered biopsies within the first year post-transplant | First year post-transplant
  total number of biopsies, indication for biopsy and CXCL10-triggered biopsies within the first year post-transplant
Safety assessed by biopsy-related complications within the first year post-transplant | First year post-transplant
  biopsy-related complications within the first year post-transplant biopsy-related complications within the first year post-transplant
Safety assessed by immunosuppression-related complications as infections and cancer within the first year post-transplant | First year post-transplant
  immunosuppression-related complications as infections and cancer within the first year post-transplant
Graft and its cause | yearly up to 10 years
  Long-term outcome Graft and its cause
Death and its cause | yearly up to 10 years
  Long-term outcome Death and its cause
Allograft function measured by creatinine and eGFR | yearly up to 10 years
  Long-term outcome Allograft function measured by creatinine and epidermal growth factor receptor (eGFR)
Proteinuria | yearly up to 10 years
  Long-term outcome Proteinuria
Biopsy-proven rejection | yearly up to 10 years
  Long-term outcome Biopsy-proven rejection

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schaub, MD, MSc, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Transplantation Immunology & Nephrology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hirt-Minkowski P, Handschin J, Stampf S, Hopfer H, Menter T, Senn L, Honger G, Wehmeier C, Amico P, Steiger J, Koller M, Dickenmann M, Schaub S. Randomized Trial to Assess the Clinical Utility of Renal Allograft Monitoring by Urine CXCL10 Chemokine. J Am Soc Nephrol. 2023 Aug 1;34(8):1456-1469. doi: 10.1681/ASN.0000000000000160. Epub 2023 May 25. PMID 37228005